CLINICAL TRIAL: NCT03772873
Title: Minimally Invasive Pilonidal Excision for the Treatment of Pilonidal Disease - A Multi-Center Non-Randomized Controlled Trial
Brief Title: MIPE for Pilonidal Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Pediatric Surgical Research Collaborative (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-0937-CCMC
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Pilonidal Disease; Pilonidal Cyst/Fistula; Pilonidal Sinus Without Abscess; Pilonidal Cyst Without Abscess; Pilonidal Cyst and Sinus Without Abscess; Pilonidal Abscess; Pilonidal Sinus With Abscess; Pilonidal Dimple With Abscess; Pilonidal Fistula With Abscess; Pilonidal Sinus Infected; Pilonidal Cyst With Sinus; Pilonidal Cyst and Sinus With Abscess; Pilonidal Disease of Natal Cleft Abscess
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIPE: Patients undergoing minimally invasive pilonidal excision with trephination.
  Interventions: Procedure: minimally invasive pilonidal excision
- Other: Patients undergoing a different procedure for pilonidal disease.

INTERVENTIONS:
Procedure: minimally invasive pilonidal excision — MIPE procedure with trephine excision of pits and sinuses
  Other Names: Gips procedure
  Groups: MIPE

SUMMARY:
Pilonidal disease often presents as a chronic, relapsing condition. A variety of procedures are used in the management of pilonidal disease, with varying degrees of morbidity, disease-free interval, and long-term success. In patients with new-onset or recurrent pilonidal disease, the investigators aim to address how minimally invasive trephine excision compares to other surgical procedures in terms of short- and long-term clinical outcomes and patient satisfaction.

In the absence of a gold standard surgical procedure, surgeon preference will help dictate the management of pilonidal disease. For many surgeons, this means a variation on open excision for pilonidal disease failing conservative management. However, outcomes for minimally invasive pilonidal excision (MIPE) as initially described by Gips and forthcoming Lipskar et al., are likely to alter management of the disease (Gips, 2008). The investigators wish to assess patient and surgeon satisfaction with MIPE, and short-term outcomes.

DETAILED DESCRIPTION:
Pilonidal disease is an inflammatory and infectious condition most often affecting young adult males. Though the pathogenesis is still debated, it is thought that tears in hair follicles of the natal cleft form small crevices where hairs and debris can collect. Over time, constant friction and stretching from daily movement pulls the debris deeper into the cavity creating a sinus. The patient is susceptible to recurrent infections because of the constant warmth, humidity, and exposure to skin and gut flora in the affected area. The clinical presentation of this condition may be acute or chronic and ranges from small, asymptomatic pits in the skin, to large abscesses with purulent and blood drainage.

Initial treatments for pilonidal disease typically include trials of conservative treatments such as improved personal hygiene with regular shaving or laser hair removal, before surgical interventions are considered. Minimally invasive options include injection of phenol, fibrin glue, cyanoacrylate into the affected areas. For patients failing conservative management, or with extensive disease, surgical management has been the standard of care.

There are a wide variety of surgical techniques for refractory pilonidal disease. These include excision with lay open or primary closure, incision and marsupialization, excision with V-Y, W-, and Z-plasty flap. Other procedures described include rhomboid excision and Limberg flap, and excision with off-midline closure. This lack of standardization suggests a complex problem without optimal treatment. The MIPE procedure with trephine excision of pits and sinuses provides an elegant solution for the majority of patients, maximizing clearance of hair follicles and diseased tissue while minimizing morbidity.

Discrepancies in recurrence rates, lengths of hospital course, time to return to work, and patients' aesthetic satisfaction between the various treatment options has led to great controversy over the best approach. Among the surgical options, some studies have reported shorter operative time, hospital stay, and time for wound healing with the excision with primary closure method, whereas flap techniques generally have a lower incidence of recurrence. However, other studies have shown shorter hospital duration and time to return to work specifically for the Limberg flap in comparison to primary closure. Controversy aside, the various surgical methods prioritize complete excision of diseased tissue at the expense of dissatisfying wound aesthetics.

MIPE with trephination was introduced by Gips et al, as an alternative excision strategy that allows for thorough pilonidal debridement while minimizing the need for general anesthesia, inpatient post-operative care, and disfiguring wound healing. Though there is an increased recurrence rate, this simple outpatient procedure allows for repeat excision at the onset of disease recurrence.

The investigators aim to study the use of this procedure in children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 25 with pilonidal disease may be included in the study. Patients with primary pilonidal disease or recurrence of pilonidal disease after previous intervention may be included.

Patients with acute pilonidal abscess or active infection may also be included in the study, provided they undergo a procedure more extensive than simple incision and drainage. At our institution, patients with acute abscess may undergo more extensive procedure at their initial operation, at surgeon discretion.

Exclusion Criteria:

* Patients who undergo simple incision and drainage for pilonidal disease as their index procedure will be excluded from the study, as this is generally a temporizing measure. Patients who undergo wide local excision, or any more complex procedure will be included within the 'standard procedure' arm. Patients who had previously undergone a simple drainage procedure and present for definitive management will be included.

Patients with significant medical comorbidities, such as cancer, diabetes mellitus, chronic steroid use, and use of immunosuppressant therapies, are excluded from the study. Any patient with an ASA III or IV will be excluded.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children presenting to clinics with symptomatic pilonidal disease and recommended for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent disease within 6 months of index surgery | 6 months
  The primary end-point will be the requirement for a second operative procedure of any kind for pilonidal disease within 6 months of initial procedure

SECONDARY OUTCOMES:
Recurrent disease within 24 months of index surgery | 24 months
  Requirement for a second operative procedure of any kind for pilonidal disease within 24 months of initial procedure
Recurrent disease within 5 years of index surgery | 5 years
  Requirement for a second operative procedure of any kind for pilonidal disease within 5 years of initial procedure
Return to school or work post procedure | 2 months
  Return to a full day of school or work following procedure
Post operative surgical site infection | 2 months
  Need for antibiotic therapy. While subjective this at least suggests a concern on the part of a healthcare provider, absent the need for objective measures such as WBC and fever.
Requirement for hospital stay | 1 week
  Any overnight stay following surgical procedure will be documented
Surgeon satisfaction with procedure | 6 months
  Surgeon questionnaire at beginning and end of enrollment on experience with procedure. Satisfaction will be measured qualitatively through a questionnaire designed for the study, detailing what procedure(s) the surgeon has performed in the past for pilonidal disease, his/her rationale for that procedure, and interest in MIPE.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Kvasnovsky, MD, PhD, MPH, Principal Investigator — Northwell Health; Abdulraouf Lamoshi, MD, Study Director — Northwell Health
Locations (10):
- United States (10):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Advocate Health Center, Park Ridge, Illinois
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Dayton Children's Hospital, Dayton, Ohio
  - Lehigh Valley Reilly Children's Hospital, Allentown, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Discussing availability of IPD with participating sites.

REFERENCES:
- [Background] Elalfy K, Emile S, Lotfy A, Youssef M, Elfeki H. Bilateral gluteal advancement flap for treatment of recurrent sacrococcygeal pilonidal disease: A prospective cohort study. Int J Surg. 2016 May;29:1-8. doi: 10.1016/j.ijsu.2016.03.006. Epub 2016 Mar 11. PMID 26975846
- [Background] Speter C, Zmora O, Nadler R, Shinhar D, Bilik R. Minimal incision as a promising technique for resection of pilonidal sinus in children. J Pediatr Surg. 2017 Sep;52(9):1484-1487. doi: 10.1016/j.jpedsurg.2017.03.040. Epub 2017 Mar 20. PMID 28366559
- [Background] Gips M, Melki Y, Salem L, Weil R, Sulkes J. Minimal surgery for pilonidal disease using trephines: description of a new technique and long-term outcomes in 1,358 patients. Dis Colon Rectum. 2008 Nov;51(11):1656-62; discussion 1662-3. doi: 10.1007/s10350-008-9329-x. Epub 2008 May 31. PMID 18516645
- [Background] Holmebakk T, Nesbakken A. Surgery for pilonidal disease. Scand J Surg. 2005;94(1):43-6. doi: 10.1177/145749690509400111. PMID 15865116